CLINICAL TRIAL: NCT04110990
Title: Retrospective Observational Study on the Epidemiological Characteristics of Influenza Patients Who Consulted in the Emergency Services of the University Hospitals of Strasbourg From September 2018 to March 2019
Brief Title: Retrospective Observational Study on the Epidemiological Characteristics of Influenza Patients
Acronym: Influenza
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7459
Record Dates: First submitted 2019-09-27; First posted 2019-10-01 (Actual); Last update posted 2019-10-02 (Actual); Status verified 2019-09

CONDITIONS: Influenza
Keywords: Influenza; Grippe; Emergency Services; Influenza, Human
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Seasonal influenza outbreaks contribute to the saturation of emergency services. Better knowledge of the epidemiology and clinical presentation of this pathology would optimize the organization of emergency reception services and provide better care for patients, disseminate educational elements to the population more appropriate as well as optimal recommendations for health professionals.

ELIGIBILITY:
Inclusion criteria:

* Major subject ((≥18 years old)
* Subject who consulted the Emergency Department of the Adult Emergencies of the Strasbourg University Hospitals between September 2018 and March 2019
* Subject for which the flu smear is positive
* Subject not expressing opposition to the use of his data for research purposes

Exclusion criteria:

* Subject having expressed his opposition to participating in the study
* Subject for which the flu smear is negative
* Subject under the protection of justice
* Subject under guardianship or curators

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient who consulted the Emergency Department of the Adult Emergencies of the Strasbourg University Hospitals between September 2018 and March 2019
Sampling Method: Non-Probability Sample
Enrollment: 384 (Estimated)
Dates: Start 2019-10 (Estimated); Primary Completion 2019-10 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Retrospectively study of the epidemiological characteristics of influenza patients consulted at the Adult Emergencies of Strasbourg University Hospitals | Files analyzed retrospectily from September 1st, 2018 to March 30, 2019 will be examined

CONTACTS AND LOCATIONS:
Overall Officials: Christine Kummerlen, MD, Study Director — University Hospital, Strasbourg, France
Locations (1):
- Service de réanimation médicale, Strasbourg, France